CLINICAL TRIAL: NCT00155428
Title: Application of Biocardiac Model in Total Correction of Tetralogy of Fallot
Brief Title: Biomodel in Tetralogy of Fallot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700518
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-05

CONDITIONS: Tetralogy of Fallot
Keywords: biomodel; rapid prototyping; computed tomograpgy
MeSH Terms: conditions — Tetralogy of Fallot

INTERVENTIONS:
Procedure: rapid prototyping
Procedure: computed tomography

SUMMARY:
Using biocardiac model in helping the total correction of the Tetralogy of Fallot.

DETAILED DESCRIPTION:
Using biocardiac model in helping the total correction of the Tetralogy of Fallot.

ELIGIBILITY:
Inclusion Criteria:

Tetralogy of Fallot

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2005-05; Study Completion 2008-12

PRIMARY OUTCOMES:
diagnostic accuracy

SECONDARY OUTCOMES:
sensitivity
specificity

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jye Chen, MD, PhD, Principal Investigator — Dept. Medical Imaging, NTUH
Locations (1):
- Dept. Medical Imaging, NTUH, Taipei, Taiwan